CLINICAL TRIAL: NCT07051057
Title: Oral Hygiene and Dietary Habits in Physical Therapy and Pharmacy Students at Sinai University
Status: Enrolling by invitation | Type: Observational
Sponsor: Sinai University (Other)
Responsible Party: Principal Investigator, Alaa Noureldeen Kora, Lecturer , Principal Investigator, Sinai University
Other Study IDs: SU.REC.2024(40H)
Record Dates: First submitted 2025-06-02; First posted 2025-07-03 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Oral Hygiene; Nutrition Habits
Keywords: Oral Hygeine; Nutrition Habits; Students; Physical Therapy; Pharamacy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Physical Therapy Group: Study the oral hygiene, nutrition habits and obesity with in the students of physical therapy Sinai university
  Interventions: Diagnostic Test: Survey using a questionnaire.
- Pharamacy Group: Study the oral hygiene, nutrition habits and obesity with in the students of the faculty of pharmacy Sinai university
  Interventions: Diagnostic Test: Survey using a questionnaire.

INTERVENTIONS:
Diagnostic Test: Survey using a questionnaire. — A survey was constructed to collect the data of oral hygiene and nutritional habits and obesity

SUMMARY:
Oral health is a multidimension domain including the human ability to talk, smile, eat, drink and swallow. Oral health has a direct relationship with the individual's quality of life and it is influenced by the perception, experiences and knowledge.

DETAILED DESCRIPTION:
Oral health is a multidimension domain including the human ability to talk, smile, eat, drink and swallow. Oral health has a direct relationship with the individual's quality of life and it is influenced by the perception, experiences and knowledge. The aim of the study is To assess the oral hygiene practices and dietary habits among physiotherapy and pharmacy students at Sinai University, To find the correlation between oral hygiene practices and dietary habits with the occurrence of oral health problems. & To compare between the oral health knowledge between physiotherapy and pharmacy students at Sinai University.

ELIGIBILITY:
Inclusion Criteria:

* A number of 334 adolescent and adults' physical therapy students at the faculty of physical therapy and 329 adolescent and adults' Pharmacy Students.
* The age from 16 to 25 years old as it is the typical age of students who are enrolled in Physical therapy and pharmacy programs.
* The subjects agreed to participate in the study, as an email address will be sent to all students that fits the criteria of selection.

Exclusion Criteria:

* Students who are enrolled to other programs rather than physical therapy and pharmacy.
* Students who are enrolled in other universities rather than Sinai university.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A number of 334 adolescent and adults' physical therapy students at the faculty of physical therapy and 329 adolescent and adults' Pharmacy Students.
Sampling Method: Non-Probability Sample
Enrollment: 663 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Oral Hygiene that students follows | "Baseline" or "Day 1"
Nutritional Habits | "Baseline" or "Day 1"

SECONDARY OUTCOMES:
Body mass index | "Baseline" or "Day 1"

CONTACTS AND LOCATIONS:
Locations (1):
- Sinai University, Ismailia, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Undecided